CLINICAL TRIAL: NCT02852057
Title: Effectiveness and Safety of Timolol and Dorzolamide Loaded Contact Lenses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201602390; OCR19613 (Other: University of Florida)
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Timolol; dorzolamide; dorzolamide-timolol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects Receiving Lenses (Experimental): All subjects who meet inclusion criteria will receive lenses loaded with timolol maleate and dorzolamide hydrochloride.
  Interventions: Drug: timolol maleate and dorzolamide hydrochloride

INTERVENTIONS:
Drug: timolol maleate and dorzolamide hydrochloride — Timolol maleate and dorzolamide hydrochloride loaded contact lenses
  Other Names: Cosopt PF

SUMMARY:
This study focuses on glaucoma therapy by drug eluting contact lenses. The contact lens will be loaded with timolol maleate and dorzolamide hydrochloride, both of which are commonly used ophthalmic drugs. Additionally, the lenses will contain vitamin E ((+) α-tocopherol) as an additive for achieving extended release of the drugs.

This study is to assess the safety of the drug loaded contact lenses and the effectiveness. Effectiveness will be a drop in IOP after using the lenses.

DETAILED DESCRIPTION:
Glaucoma is the second largest cause of blindness in the world (largest amongst African-Americans) and affects about 66.8 million people, leaving 6.7 million with bilateral blindness. The World Health Organization estimates that by 2020 the number of cases for blindness due to glaucoma will double to 12 million. The financial impact of glaucoma on the US economy is more than $1.5 billion annually.

Glaucoma can be managed through several intra ocular pressure (IOP) lowering medications including Pfizer's XALATAN® (latanoprost), which accounted for 27% of the total US market in Jan 2010. Effective management however requires patient-compliance, which is frequently low for eye drop based therapies. The compliance is less than 50% for glaucoma eye drops, and even lower for multiple drops and/or multiple drug therapies. In a recent study with 204 glaucoma patients, only 71% were able to instill the drop into the eye, with only 39% doing it without touching the bottle to the eye surface. The lack of patient-compliance to glaucoma therapy arises from several sources. Firstly, due to the chronic nature of the disease, patients on glaucoma medication cannot immediately discern the benefits of taking the medication regularly, and so they are not sufficiently motivated to be compliant. Even for patients that regularly take the medicine through eye drops, the compliance can be far from perfect due to the difficulties in instilling eye drops.

In addition to the lack of compliance, low bioavailability of glaucoma drugs delivered through eye drops is a major problem, which can lead to side effects ranging from irritation and the unpleasant taste to debilitating effects such as heart problems. The corneal bioavailability of glaucoma drugs ranges in 1-5% because of the rapid tear turn over accompanied by drug transport into the conjunctiva, which has a larger area and permeability compared to cornea. The conjunctival and nasal absorption leads to systemic exposure in all tissues, and thus leading to potential side effects. The presence of preservatives such as benzalkonium chloride (BAK) further contributes to toxicity from eye drops.

The deficiencies of the eye drop formulations for glaucoma therapy were addressed by Ocusert® (Alza), a highly successful pilocarpine releasing ocular insert that was placed in the cul de sac of the eye. Ocusert® was shown in clinical studies to produce a constant reduction in IOP for over 7 days 23. The total dosage of pilocarpine administered by one Ocusert® system over 7-days was about one-eighth of the amount provided by the 28 applications (4 each day) of the 2% eyedrops. The simplified regimen and reduced side effects from Ocusert® encouraged patient compliance. Unfortunately, the manufacturer of Ocusert® has discontinued making them likely due to some drawbacks of the device including retention problems, twisting to change shape, sight impediment due to dislocation of the device in front of the pupil, but most important a sudden burst release in 0.4% of cases that could cause toxicity. Additionally, pilocarpine has been replaced by several newer drugs such as prostaglandins as the first line of defense against glaucoma. Our goal in this proposed research is to replicate the success of Ocusert® with a newer drug and a different device design to eliminate the drawbacks of Ocusert®. To improve compliance and reduce side effects, we propose to develop a drug delivery system that has excellent retention and biocompatibility, with continuous release of drugs for extended durations, with high bioavailability and with no possibility of drug leakage.

Contact lenses have the highest possible bioavailability for cornea because drug released by contact lenses is trapped in the thin post lens tear film between the cornea and the lens for extended period longer than 30 minutes, compared to 2-5 minutes for eye drops. The increased residence time leads to very high fractional drug uptake by cornea, which reduces the needed dose, thereby improving the safety profile. The use of contact lenses for treating glaucoma will also result in very high compliance for the patients who also need vision correction because they will always insert the lens for the vision correction, even if they do not immediately appreciate the benefits of the IOP reduction. Additional benefits of contact lens based drug delivery will be elimination of the preservatives in the multi-use eye drop formulations, which can cause discomfort and redness. Finally, contact lenses are the most commonly used medical devices with over 41 million wearers in the United States and over five decades of history of safe use. Based on all these considerations, drug loaded contact lenses could be very promising for delivery of ophthalmic drugs.

ELIGIBILITY:
Inclusion Criteria:

1. At baseline visit IOP > 18 mm Hg and < 35 mm Hg, with difference between eyes of < 5 mm Hg
2. Willingness to participate in washout period and to wear glasses if necessary
3. Corneal thickness between 480 and 620 microns
4. Shaffer Angle > 2
5. Visual acuity of 20/200 or better
6. Binocular
7. Age 18 or over and willing and able to give consent

Exclusion Criteria:

1. Pregnancy
2. Asthma
3. Bradycardia
4. Steven's Johnson
5. Sulpha drug intolerance
6. Corneal ulcers or other corneal complications
7. Dry eyes requiring two or more instillation of rewetting drops per day
8. Any previous incidence of contact lens intolerance
9. Highly aspheric cornea that would make fitting a contact lens difficult (i.e., keratoconus)
10. Participation in any drug clinical trial in the last three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
IOP | Day 1, Day 2, Day 4, Day 7, and Day 9
  Pressure will be measured in trial subjects before placement of lenses and after day 1, day 2, day 4, day 7, and day 9

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sherwood, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States